CLINICAL TRIAL: NCT00431613
Title: Sequential Administration of Docetaxel/Gemcitabine Followed by Concurrent Chemo-radiotherapy, With or Without Consolidation Chemotherapy, as First Line Treatment in Patients With Unresectable Stage IIIA/IIIB NSCLC. A Randomized Phase II Study
Brief Title: Study of Docetaxel/Gemcitabine Followed by Chemo-radiotherapy (Chemo-RT), With or Without Consolidation Chemotherapy, in IIIA/IIIB Non Small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to Poor Accrual
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/04.26
Record Dates: First submitted 2007-02-05; First posted 2007-02-06 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; Induction chemotherapy; Concurrent chemoradiotherapy; Consolidation therapy; Docetaxel; Gemcitabine; Carboplatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Gemcitabine; Carboplatin; Chemoradiotherapy

ARMS (2):
- 1 (Experimental): DG -> RT
  Interventions: Drug: Docetaxel; Drug: Gemcitabine; Radiation: Chemoradiotherapy
- 2 (Experimental): DG -> RT -> DCarbo
  Interventions: Drug: Docetaxel; Drug: Gemcitabine; Drug: Carboplatin; Radiation: Chemoradiotherapy

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 75 mg/m2 IV on day 8 every 3 weeks for 2 cycles
  Other Names: Taxotere
Drug: Gemcitabine — Gemcitabine 1100 mg/m2 on days 1 and 8 every 3 weeks for 2 cycles
  Other Names: Gemzar
Drug: Carboplatin — Carboplatin 6AUC IV on day 1 every 3 weeks for 3 cycles
  Arms: 2
Radiation: Chemoradiotherapy — After 21 days from the 2nd chemotherapy cycle definitive concurrent chemoradiotherapy will be started: daily fractions of 1.8 Gy for 5 days/week, for a total dose of 45 Gy.
  During the radiotherapy docetaxel 25 mg/m2, IV, will be administered on days 1, 8, 15, 22, 29 and carboplatin 2AUC, IV , on days 4, 11, 18, 25, 32
Drug: Docetaxel — Docetaxel 75mg/m2 IV on day 1 for 3 cycles
  Other Names: Taxotere
  Arms: 2

SUMMARY:
The combination of chemotherapy with radiotherapy remains the standard of therapy for patients with stage III NSCLC. A recent phase II study has presented encouraging data regarding the administration of docetaxel as consolidation treatment after definitive concurrent chemo-radiotherapy.

DETAILED DESCRIPTION:
To evaluate whether the administration of consolidation therapy with docetaxel/carboplatin after induction chemotherapy followed by concurrent chemoradiotherapy, offers any advantage regarding time to tumor progression

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed, unresectable locally advanced (stage IIIA/IIIB) NSCLC
* no previous therapy for NSCLC is allowed
* age >18 years
* bidimensionally measurable disease
* performance status (WHO) 0-2
* absence of pleural effusion
* adequate liver (serum bilirubin < 1.5 times the upper normal limit (UNL); AST and ALT < 2.5 times the UNL in the absence of demonstrable liver metastases, or < 5 times the UNL in the presence of liver metastases); adequate renal function (serum creatinine < 1.5 times the UNL); and bone marrow (neutrophils ≥ 1.5x 109 /L, and platelets ≥ 100x 109 /L) function
* life expectancy of more than 3 months
* written informed consent

Exclusion Criteria:

* active infection
* history of significant cardiac disease (unstable angina, congestive heart failure, myocardial infarction within the previous 6 months, ventricular arrhythmias)
* malnutrition (loss of ≥ 20% of the original body weight)
* performance status: 3-4
* sensor or motor neuropathy > grade I
* second primary malignancy, except for non-melanoma skin cancer
* psychiatric illness or social situation that would preclude study compliance
* pregnant or lactating women

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-03; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Time to tumor progression (TTP) | 1 year

SECONDARY OUTCOMES:
Response rate | Objective responses confirmed by CT or MRI (on 3rd and 6th cycle)
Overall survival | Probability of 1-year survival (%)
Toxicity | Toxicity assessment on each chemotherapy cycle
Quality of life | Assessment every two cycles
Symptom improvement | Assessment every two cycles

CONTACTS AND LOCATIONS:
Overall Officials: Vassilis Georgoulias, MD, Principal Investigator — University Hospital of Crete
Locations (10):
- Greece (10):
  - University Hospital of Crete, Heraklion, Crete
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - 401 Military Hospital, Medical Oncology Unit, Athens
  - Air Forces Military Hospital, Dep of Medical Oncology, Athens
  - IASO General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - Laikon General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - Sismanogleio General Hospital, 1st, 2nd Dep of Pulmonary Diseases, Athens
  - Sotiria General Hospital, 1st, 3rd, 6th, 7th, 8th Dep of Pulmonary Diseases, Athens
  - Metaxa's Anticancer Hospital of Piraeus,1st Dep of Medical Oncology, Piraeus
  - Theagenion Anticancer Hospital of Thessaloniki, Thessaloniki